CLINICAL TRIAL: NCT05730296
Title: The Effects of Repetitive Transcranial Magnetic Stimulation in Older Adults With Mild Cognitive Impairment - Randomized Controlled Study
Brief Title: Transcranial Magnetic Stimulation in Patients With Mild Cognitive Impairment - RCT Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUBZ.C230.22.062.TMS.MCI
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment
Keywords: rTMS, MCI, TMS, RCT
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): rTMS active + training
  Interventions: Device: TMS
- group 2 (Experimental): rTMS active
  Interventions: Device: TMS
- sham coil (Sham Comparator): rTMS sham
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — 10 rTMS sessions combined with cognitive training
  Arms: group 1
Device: TMS — 10 rTMS sessions
  Arms: group 2
Device: TMS — 10 sham coils sessions without cognitive training
  Arms: sham coil

SUMMARY:
The study is planned as a randomized, double-blind, and sham-controlled parallel trial, in which raters and participants will be blinded to the group selection. A total of 60 participants, meeting the eligibility criteria, will be enrolled in the study and divided randomly into 3 groups (2 experimental ones with active rTMS, one of which with the addition of cognitive training RehaCom, one control group with sham-placebo rTMS).

DETAILED DESCRIPTION:
The study is planned as a randomized, double-blind, and sham-controlled parallel trial, in which raters and participants will be blinded to the group selection. A total of 60 participants, meeting the eligibility criteria, will be enrolled in the study and divided randomly into 3 groups (2 experimental ones with active rTMS, with and without the addition of cognitive training RehaCom, one control group with sham-placebo rTMS).

Experimental group 1 (E1, n=20): patients undergoing rTMS and computerized cognitive training Experimental group 2 (E2, n=20) patients undergoing TMS without training of cognitive function Control group (CG, n=20) - patients with placebo TMS - sham coil without cognitive training

The following stimulation protocol will be used to conduct research into the treatment of mild cognitive impairment.

The target area in rTMS is the dorsolateral prefrontal cortex of the left hemisphere of the brain, mostly responsible for operational memory, memory of everyday events, information processing and learning. Delivering rTMS protocol is characterized by two thousand pulses at 10 Hz, 5-s train duration, and 25-seconds intervals at 110% of motor threshold five times a week for two weeks. The following protocol has been chosen based on reports from the article by Hellen Livia Drumond et at. (2015). In this study the research group has demonstrated that after 10 sessions of active TMS (two thousand pulses at 10 Hz, 5-s train duration, and 25-seconds intervals at 110% of motor threshold five times a week for two weeks) crucial for MCI cognitive domains such as episodic memory and logical memory.

ELIGIBILITY:
Detailed inclusion Criteria:

* participants of both sexes with MCI
* informed consent to undergo rTMS and study protocol

Screening procedure of cognitive deficits:

* confirmation of the diagnosis of MCI according to Petersen's criteria (concern related to the change in cognitive performance, deterioration in one or more cognitive areas, maintaining the independent ability of daily functioning, lack of dementia)
* confirmation of the diagnosis of MCI based on the results obtained in neuropsychological tests (MoCA, Montreal Cognitive Assessment test and CDR, Clinical Dementia Rate)

Detailed exclusion criteria (TMS and fMRI)

Contraindications to treatments using TMS:

* positive history of epileptic seizures or a positive family history of epilepsy
* magnetic or ferromagnetic implants, both electronic (e.g., heart/brain stimulators) as well as mechanical (eg bone anastomoses) within the head and neck
* previous stroke or head injury with identified neurological deficits
* increased intracranial pressure or a positive history of increased intracranial pressure
* pregnant women and women during lactation

Contraindications to MR examinations:

* claustrophobia
* magnetic or ferromagnetic implants, both electronic (e.g., cardiac/brain stimulators) as well as mechanical (eg bone anastomoses) within the head and neck
* other psychiatric disorders (i.e. depression, anxiety disorders), which may affect cognitive performance (GDS-15, 15-Item Geriatric Depression Scale; HAMA-14, 14-Item Hamilton Anxiety Scale)
* braces
* occurrence of significant pathologies in the cerebrum area (tumors, hydrocephalus, strokes)
* lack of patient's informed consent
* documented persistent lack of cooperation in treatment

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of efficiency of rTMS active and sham-placebo stimulation Change from baseline to END of stimulation regarded as reduction of symptoms of cognitive disorders measured by CANTAB test | END of stimulation
  Comparison of efficiency of rTMS active and rTMS sham placebo stimulation from baseline to end of stimulation measured with The Cambridge Neuropsychological Test Automated Battery (CANTAB). The CANTAB includes highly sensitive, precise and objective measures of cognitive function, correlated to neural networks with demonstrated sensitivity to detecting changes in neuropsychological performance. The battery includes tests of working memory, learning and executive function; visual, verbal and episodic memory; attention, information processing and reaction time; social and emotion recognition, decision making and response control.Cognitive performance testing using selected CANTAB will examine: attention (Reaction Time test), visual memory (Paired Association Learning, Pattern Recognition Memory), executive functions and operating memory (Spatial Working Memory).
Comparison of efficiency of rTMS active and sham-placebo stimulation Change from baseline to END of stimulation regarded as reduction of symptoms of cognitive disorders measured by FAS test | END of stimulation
  Comparison of efficiency of rTMS active and rTMS sham placebo stimulation from baseline to end of stimulation measured by verbal fluency FAS test. Verbal fluency is measured by requesting an individual to orally produce as many words as possible that begin with the letters F, A, and S within a prescribed time frame (1 minute in the research).
Comparison of efficiency of rTMS active and sham-placebo stimulation Change from baseline to END of stimulation regarded as reduction of symptoms of cognitive disorders measured by DemTect test. | END of stimulation
  Comparison of efficiency of rTMS active and rTMS sham placebo stimulation from baseline to end of stimulation measured by DemTect scale. DemTect is a screening test for MCI and early stages of dementia, especially sensitive to memory deficits. The whole test consists of 5 subscales: (1) a word list, (2) number transcoding, (3) supermarket (semantic fluency), (4) digit span reverse and (5) word list delayed recall.
Comparison of efficiency of rTMS active and rTMS sham placebo stimulation from baseline to end of stimulation measured by neuroimaging parameters derived from volumetry, DTI and rs fMRI. | END of stimulation
  Comparison of efficiency of rTMS active and rTMS sham placebo stimulation from baseline to end of stimulation measured by neuroimaging parameters derived from volumetry, DTI and rs fMRI. Brain MRI will be performed with a 3 Tesla (Ingenia, Philips Best) scanner using standard anatomical sequences include the following high resolution sequences: 3D T1-weighted, 3D-T2-weighted, 3D Flair and post gadolinium 3DT1-weighted imaging followed by new advanced techniques such as brain volumetry, DTI and rs-fMRI. All participants will undergo brain standard MR imaging using a 32-channel coil dedicated for head examination before and after rTMS.

SECONDARY OUTCOMES:
Comparison of efficiency of rTMS active and sham-placebo stimulation Change from baseline to END of stimulation regarded as reduction of symptoms of apathy measured by AES scale. | END of stimulation
  Comparison of efficiency of rTMS active and sham-placebo stimulation Change from baseline to END of stimulation regarded as reduction of symptoms of apathy measured by Apathy Evaluation Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Rymaszewska, Professor, Study Director — Wroclaw Medical Univeristy, Department of Psychiatry
Locations (1):
- Wroclaw Medical University, Department of Psychiatry, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No